CLINICAL TRIAL: NCT01835951
Title: Individual Versus Grouped Debriefing Approaches in Anaesthesia Crisis Simulation-Based Training. What Impact On The Technical Score ?
Acronym: DEBRIEF-SIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Floriane CICERON, Anesthesia-reanimation internal, Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EI/2012/028
Record Dates: First submitted 2013-03-29; First posted 2013-04-19 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Cardiac Arrest; Pregnancy
Keywords: Simulation; Debriefing; Anaesthesia Crisis Management; Cardiac Arrest; Pregnancy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual Debriefing (Other): Individual debriefing consists in a individual meeting between each subject of the study and the investigator to analyze the management of the anaesthesia crisis simulated.
  Interventions: Other: Individual Debriefing
- Grouped Debriefing (Other): Grouped debriefing consists in the analysis of the management of the anaesthesia crisis simulated in the presence of all the subject included in the Grouped Debriefing group.
  Interventions: Other: Grouped Debriefing

INTERVENTIONS:
Other: Grouped Debriefing — Debriefing consists in an analysis by the investigator of the management of the anaesthesia crisis simulated in the presence of all the subjects included in the Groupe Debriefing group.
  Arms: Grouped Debriefing
Other: Individual Debriefing — Individual debriefing consists in a individual meeting between each subject of the study and the investigator to analyze the management of the anaesthesia crisis simulated.
  Arms: Individual Debriefing

SUMMARY:
Simulation-based training is essential in learning or maintaining skills in high risk industry such as aviation and railway and in the medical field like anaesthesia. Debriefing following simulation is fundamental in order to reduce the emotional impact of the session and to asses the technical and non-technical skills (behavior). Even if the ideal debriefing method is still to be found, individual debriefing is considered as the gold standard but time consuming. The DEBRIEF-SIM study is a prospective, single blinded, multicentric and randomized study that will compare the individual (defined by learning couple resident and nurse) approach to a grouped (several couples) debriefing. The primary end point is to define the noninferiority of this approach compared to the individual one on the educational impact.

The learners will be debriefed according to their randomization after the first session, but will all undergo individual debriefing following the second session.

DETAILED DESCRIPTION:
Individual debriefing consists in a individual meeting between each subject of the study and the investigator to analyze the management of the anaesthesia crisis simulated.

Grouped debriefing consists in the analysis by the investigator of the management of the anaesthesia crisis simulated in the presence of all the subjects included in the Grouped Debriefing group.

ELIGIBILITY:
Inclusion Criteria:

* Doctor:

  * resident in anesthesia and intensive care CHU Besançon and Dijon

Student nurse anesthetist:

* Student nurse anesthesist 1st or 2nd year of school Besançon and Dijon

Exclusion Criteria:

* Subjects incapable of giving consent: incapacitated (subjects under guardianship), minors (< 18 years)
* Refusal to participate in the study
* Refusal to sign the confidentiality clause

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Score of technical competence | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Pili-Floury, Principal Investigator — Faculté de Franche-Comté des Etudes de Médecine et Pharmaceutiques
Locations (1):
- Faculté de Franche-Comte des études de medecine et pharmaceutiques, Besançon, France